CLINICAL TRIAL: NCT02975375
Title: The Impact of Perioperative Geriatric Care on Outcomes After Elective Noncardiac Surgery
Status: Completed | Type: Observational
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: DM4
Record Dates: First submitted 2016-11-17; First posted 2016-11-29 (Estimated); Results first posted 2025-03-17 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-02

CONDITIONS: SURGICAL PROCEDURES, OPERATIVE; Aged; Epidemiology; Mortality
MeSH Terms: interventions — Restraint, Physical

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Preoperative geriatric consult or assessment: Patients who have a geriatric assessment of consult billed in the 4 months before surgery
  Interventions: Procedure: Preoperative geriatric consult or assessment
- No Preoperative geriatric consult or assessment: Patients who do not have a geriatric assessment of consult billed in the 4 months before surgery
  Interventions: Procedure: No Preoperative geriatric consult or assessment

INTERVENTIONS:
Procedure: Preoperative geriatric consult or assessment — A preoperative geriatric consult or assessment will be considered to be present if such a consult or assessment is billed by a geriatrician for a patient in the cohort within 4 months preceding surgery. For the primary analysis we will collapse both geriatric consultations and comprehensive geriatric assessments into a single exposure level.
  Groups: Preoperative geriatric consult or assessment
Procedure: No Preoperative geriatric consult or assessment — No assessment or consult billed in the 4 months before surgery
  Groups: No Preoperative geriatric consult or assessment

SUMMARY:
The investigators will conduct a population-based study using health administrative data to evaluate the impact of preoperative geriatric consultation on postoperative outcomes in older patients having elective, non-cardiac surgery

DETAILED DESCRIPTION:
The investigators will use multilevel multivariable analyses to measure the association between preoperative geriatric assessment or consultation and outcomes after major elective non-cardiac surgery. Sensitivity analyses will be done to evaluate types and timing of geriatric care around surgery, as well as for effect modification based on patient and procedural factors.

ELIGIBILITY:
Inclusion Criteria:

* >65
* Resident of Ontario
* Having elective non-cardiac surgery (inpatient admission)

Exclusion Criteria:

* Residing in a nursing home or long term care facility at baseline

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Individuals >65 years of age on the day of the potential participant's first elective non-cardiac surgery in the study period
Sampling Method: Non-Probability Sample
Enrollment: 266499 (Actual)
Dates: Start 2002-04; Primary Completion 2014-03 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Ottawa Hospital Research Institute, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Preoperative Geriatric Consult or Assessment | No Preoperative Geriatric Consult or Assessment
Started | 7352 | 259147
Completed | 7352 | 259147
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Preoperative Geriatric Consult or Assessment | No Preoperative Geriatric Consult or Assessment | Total
Number analyzed (Participants) | 7352 | 259147 | 266499
Age, Continuous [Mean (Standard Deviation); unit: years] | 75.0 (6.3) | 74.2 (6.2) | 74.6 (6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4400 | 137096 | 141496
  Male | 2952 | 122051 | 125003
Neighbourhood Income Quintile [Median (Inter-Quartile Range); unit: Neighbourhood income quintile] — Neighborhood socioeconomic status of the participants is presented as income quintile (income quintile is a measure of neighbourhood socioeconomic status that divides the population into five income groups (from lowest income to highest income)). The scale is from 1-5 (income group quintile 1 (lowest), 2, 3, 4, 5 (highest)). The groups are based on where 20% of the population falls within each category and therefore values vary by year.
  Neighbourhood income quintile | 3 [4 to 5] | 3 [4 to 5] | 3 [4 to 5]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With All-Cause Mortality at 90-days
Description: Death from any cause in the 90 days after surgery
Time Frame: date of surgery to 90 days after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Preoperative Geriatric Consult or Assessment | No Preoperative Geriatric Consult or Assessment
Number analyzed (Participants) | 7352 | 259147
Participants | 103 | 6172

2. Secondary Outcome: Patient Safety Event
Description: Any Type 2 diagnostic code for a patient-safety event
Time Frame: From surgery to hospital discharge (on average 6 to 7 days)
Measure: Count of Participants; unit: Participants
Arm/Group | Preoperative Geriatric Consult or Assessment | No Preoperative Geriatric Consult or Assessment
Number analyzed (Participants) | 7352 | 259147
Participants | 1129 | 50256

3. Secondary Outcome: Hospital Length of Stay
Time Frame: date of surgery to date of hospital discharge, or 365 days after surgery, whichever comes first
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Preoperative Geriatric Consult or Assessment | No Preoperative Geriatric Consult or Assessment
Number analyzed (Participants) | 7352 | 259147
Days | 6.0 (7.3) | 7.1 (10.3)

4. Secondary Outcome: Non-independent Discharge Location
Description: Discharge disposition from hospital record that is not a home discharge without support
Time Frame: date of surgery to date of hospital discharge, or 365 days after surgery, whichever comes first
Measure: Count of Participants; unit: Participants
Arm/Group | Preoperative Geriatric Consult or Assessment | No Preoperative Geriatric Consult or Assessment
Number analyzed (Participants) | 7352 | 259147
Participants | 5264 | 145822

5. Secondary Outcome: 30-day Hospital Readmission
Description: New acute care hospitalization within 30-days of discharge from the index hospitalization
Time Frame: Date of discharge (on average 6 to 7 days) to 30 days after discharge (on average 5 weeks)
Measure: Count of Participants; unit: Participants
Arm/Group | Preoperative Geriatric Consult or Assessment | No Preoperative Geriatric Consult or Assessment
Number analyzed (Participants) | 7352 | 259147
Participants | 643 | 20656

ADVERSE EVENTS:
Time Frame: 90 Days
Description: All cause mortality: the occurrence of death due to any cause was collected. No other adverse events were collected.
Arm/Group | Preoperative Geriatric Consult or Assessment | No Preoperative Geriatric Consult or Assessment
All-Cause Mortality (participants affected / at risk) | 103/7352 | 6172/259147
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
This was an observational study, so we cannot prove causality. Unmeasured confounding is a risk to causal inference, but we were able to control for a large number of confounders, including mortality risk, diagnoses, preoperative healthcare use, and unmeasured hospital-level confounders. We were unable to study all possible pathways, such as improvements in medication appropriateness, that may be attributable to geriatric care.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No